CLINICAL TRIAL: NCT00354900
Title: Phase I Study of Aprotinin in Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The FDA changed the labeling for this agent, and we felt we could not offer it to patients on a non-surgical study.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0540
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; fibrinolysis; urokinase-type plasminogen activator; plasminogen activator inhibitor; aprotinin; plasmin/alpha-2-antiplasmin complex
MeSH Terms: conditions — Breast Neoplasms | interventions — Aprotinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aprotinin

SUMMARY:
There is an intimate relationship between processes which promote growth, invasion, and metastasis of cancers, and processes which regulate blood clotting. The enzymes uPA and PAI-1 are key regulators of the remodeling of recently formed blood clots, and there is substantial information linking greater levels of uPA and PAI-1 in breast cancers with a greater likelihood of breast cancer recurrence and death. As uPA and PAI-1 are excellent markers for a cancer's aggressive clinical behavior, uPA and PAI-1 may be potential targets for anticancer therapy. Aprotinin is an inhibitor of uPA activation, and has been approved by the FDA to reduce blood loss in patients undergoing cardiopulmonary bypass surgery. Studies in animals and limited studies in patients have shown that Aprotinin slows the growth of tumors. Our hypothesis is that uPA is chronically activated in malignancies, and that inhibition of uPA by Aprotinin would slow the rate of progression of breast cancer.

DETAILED DESCRIPTION:
Urokinase-type plasminogen activator (uPA) is a serine protease whose physiologic function is to catalyze the conversion of plasminogen to the active proteolytic form, plasmin, for participation in processes which require tissue remodeling such as wound healing, embryogenesis and inflammatory responses. uPA is among numerous tissue proteases also found in association with neoplastic disease, playing a pathologic role in tumor growth and metastasis. The activity of uPA can be neutralized by a specific inhibitor, plasminogen activator inhibitor type-1 (PAI-1) which forms inactive complexes of 1:1 stoichiometry with the plasminogen activators. Through inhibition of uPA and tPA, PAI-1 inhibits plasmin; the inhibitory effect should limit the extent of extracellular matrix protein degradation and reduce activation of MMP's and angiogenic growth factors such as VEGF. However, tissue overexpression of PAI-1 correlates with more aggressive clinical behavior of the malignancy. In fact, the upregulation of PAI-1 may be a cellular attempt to return to homeostasis, which is disrupted by activation of uPA or other factors. Upregulation of PAI-1 may be an indicator that uPA or some other pathway is contributing to an aggressive phenotype. Co-expression of uPA and PAI-1 in primary breast tumor tissue is associated with a greater risk of locoregional and distant recurrence, a poorer response to adjuvant hormonal or chemotherapy, and a shorter survival. Elevation of circulating PAI-1 in patients with metastatic breast cancer is associated with a shorter survival.

We hypothesize that uPA activation is in part responsible for the clinical progression of malignancy. Inhibition of uPA is therefore a rational strategy for the control of advanced breast cancer. Aprotinin is a safe and effective protease inhibitor of both uPA and plasmin. Aprotinin is approved for the treatment of septic shock, and for the prevention of blood loss in patients undergoing cardiopulmonary bypass surgery. In patients undergoing cardiopulmonary bypass surgery, Aprotinin blunts the acute increase in fibrinolytic activity caused by uPA, and decreases the expression of counter-regulatory PAI-1. In several in vivo tumor models, Aprotinin inhibits tumor growth, invasiveness, and metastasis. Limited experience in patients with cancer suggests prolongation of survival in patients treated with a single or multiple doses of Aprotinin. We hypothesize that Aprotinin would delay disease progression by decreasing the chronic activation of uPA and PAI-1, and that delay of tumor progression would correlate with inhibition of laboratory measures of fibrinolysis.

This is a Phase I trial. Patients with metastatic breast cancer will receive escalating doses of Aprotinin in one of four dose cohorts, ranging from 2.0 x 106 KIU to 6.0 x 106 KIU. Three to six patients will be entered at each dose cohort, and the maximum tolerated dose will be defined as the highest dose at which fewer than 33% of patients experience a dose limiting toxicity. A total of nine patients will be entered at the maximum tolerated dose. The extent of disease will be assessed radiologically at baseline, and again at 6, 12, 18, and 24 weeks after treatment with Aprotinin. Coagulation parameters, including PT/PTT, D-Dimer, FDP's, uPA, and PAI-1 will be assayed at baseline, and at several intervals out to 30 days after treatment with Aprotinin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically proven metastatic breast cancer.
* Patients with at least one bidimensionally measurable lesion (diameter > 1 cm), or an evaluable bone lesion that will not undergo biopsy.
* Age > 18 years.
* Life expectancy of at least 6 months.
* ECOG performance status 0-3.
* Screening laboratories within the following parameters: ANC > 1500 cells/mm3, Platelets > 100,000 cells/mm3, AST < 2 x upper limit of normal, Bilirubin < 1.5 x upper limit of normal, Calculated creatinine clearance > 30 cc/min by the Cockroft and Gault equation.
* Concurrent treatment with hormonal therapy or trastuzumab is allowed.
* Patients must be post-menopausal (either as a result of surgery, or amenorrhea for at least 12 consecutive months), or they must be practicing either abstinence, an adequate method of contraception (intrauterine device or barrier contraception), or their sexual partner must be sterile. Women who are pregnant, breast-feeding, or who are fertile and not practicing an adequate means of contraception will be excluded.
* Patients must have a central venous catheter.
* Patients must be able to give informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

* No known CNS metastases.
* No treatment with cytotoxic chemotherapy allowed within 21 days of treatment with Aprotinin.
* No treatment with investigational agents allowed within 21 days of treatment with Aprotinin.
* No severe cardiovascular disease including unstable heart rhythm, uncompensated congestive heart failure, unstable angina or myocardial infarction within 6 months.
* No bleeding diathesis or coagulopathy including concomitant use of anticoagulants for thromboembolic disease
* No active anticoagulant therapy (including antiplatelet agents) for at least ten days.
* No active, uncontrolled bacterial, viral or fungal infection.
* No patients who are known or expected to be allergic to aprotinin, or who have received prior aprotinin.
* No patient with chronic systolic blood pressure (SBP) < 90 mm Hg. If the (SBP) is < 90 mm Hg on the day of treatment intravenous fluid may be administered to restore intravascular volume, if clinically indicated. In such case, if IV fluid corrects the SBP then the study drug may be given

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-07; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated single dose of Aprotinin in patients with advanced breast cancer

SECONDARY OUTCOMES:
To determine the toxicities of a single infusion of Aprotinin in patients with advanced breast cancer
To determine the progression free survival and overall survival following a single dose of Aprotinin in patients with advanced breast cancer
To determine the effects of a single dose of Aprotinin on markers of the coagulation pathway

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Schwartz, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States